CLINICAL TRIAL: NCT00574496
Title: An Intention-to-Treat Study of Salvage Chemotherapy Followed by Allogeneic Hematopoietic Stem Cell Transplant for the Treatment of High-Risk or Relapsed Hodgkin Lymphoma
Brief Title: Combination Chemotherapy Followed by Donor Stem Cell Transplant in Treating Patients With Relapsed or High-Risk Primary Refractory Hodgkin Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-147; MSKCC-07147
Record Dates: First submitted 2007-12-14; First posted 2007-12-17 (Estimated); Results first posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2022-10

CONDITIONS: Lymphoma
Keywords: recurrent adult Hodgkin lymphoma; recurrent/refractory childhood Hodgkin lymphoma; adult lymphocyte depletion Hodgkin lymphoma; adult nodular sclerosis Hodgkin lymphoma; adult mixed cellularity Hodgkin lymphoma; childhood lymphocyte depletion Hodgkin lymphoma; childhood mixed cellularity Hodgkin lymphoma; childhood nodular sclerosis Hodgkin lymphoma; stage III adult Hodgkin lymphoma; stage IV adult Hodgkin lymphoma; stage III childhood Hodgkin lymphoma; stage IV childhood Hodgkin lymphoma
MeSH Terms: conditions — Lymphoma; Hodgkin Disease; Recurrence | interventions — Cyclophosphamide; Cyclosporine; fludarabine phosphate; Gemcitabine; Ifosfamide; Mechlorethamine; Melphalan; Methotrexate; Mycophenolic Acid; Prednisone; Procarbazine; Vincristine; Vinorelbine; Peripheral Blood Stem Cell Transplantation; Cord Blood Stem Cell Transplantation; Whole-Body Irradiation

ARMS (1):
- High-Risk or Relapsed Hodgkin Lymphoma (Experimental): This is a phase 2 intention-to-treat study of salvage chemotherapy followed by allogeneic HSC transplant for the treatment of primary refractory or relapsed HL. Patients who 1) do not progress on salvage chemotherapy, and 2) have both suitable HSC donors and 3) a satisfactory pre-allograft work-up will proceed to allograft. Patients who fail any of these 3 criteria will be off-study and considered treatment failures for the purposes of the intention-to-treat study.
  Interventions: Drug: cyclophosphamide; Drug: cyclosporine; Drug: fludarabine phosphate; Drug: gemcitabine hydrochloride; Drug: ifosfamide; Drug: mechlorethamine hydrochloride; Drug: melphalan; Drug: methotrexate; Drug: mycophenolate mofetil; Drug: prednisone; Drug: procarbazine hydrochloride; Drug: vincristine sulfate; Drug: vinorelbine tartrate; Procedure: allogeneic bone marrow transplantation; Procedure: allogeneic hematopoietic stem cell transplantation; Procedure: nonmyeloablative allogeneic hematopoietic stem cell transplantation; Procedure: peripheral blood stem cell transplantation; Procedure: umbilical cord blood transplantation; Radiation: total-body irradiation

INTERVENTIONS:
Drug: cyclophosphamide
Drug: cyclosporine
Drug: fludarabine phosphate
Drug: gemcitabine hydrochloride
Drug: ifosfamide
Drug: mechlorethamine hydrochloride
Drug: melphalan
Drug: methotrexate
Drug: mycophenolate mofetil
Drug: prednisone
Drug: procarbazine hydrochloride
Drug: vincristine sulfate
Drug: vinorelbine tartrate
Procedure: allogeneic bone marrow transplantation
Procedure: allogeneic hematopoietic stem cell transplantation
Procedure: nonmyeloablative allogeneic hematopoietic stem cell transplantation
Procedure: peripheral blood stem cell transplantation
Procedure: umbilical cord blood transplantation
Radiation: total-body irradiation

SUMMARY:
RATIONALE: Giving chemotherapy before a donor stem cell transplant helps stop the growth of cancer cells. It also helps stop the patient's immune system from rejecting the donor's stem cells. When the healthy stem cells from a donor are infused into the patient they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets. Sometimes the transplanted cells from a donor can make an immune response against the body's normal cells. Giving cyclosporine, mycophenolate mofetil, and methotrexate before and after transplant may stop this from happening.

PURPOSE: This phase II trial is studying how well combination chemotherapy followed by donor stem cell transplant works in treating patients with relapsed or high-risk primary refractory Hodgkin lymphoma.

DETAILED DESCRIPTION:
OUTLINE: Patients are stratified according to response to prior therapy and risk factors (those with presence of all 3 risk factors and failed primary therapy or primary progressive disease vs. patients who relapse more than 100 days after an autologous stem cell transplant).

* Salvage chemotherapy (IGV or MOPP): Patients who have previously received mechlorethamine hydrochloride receive IGV; patients who have previously received a gemcitabine-based regimen receive MOPP.

  * IGV (ifosfamide, gemcitabine hydrochloride, and vinorelbine ditartrate): Patients receive IGV combination chemotherapy comprising ifosfamide IV on days 1-4, gemcitabine hydrochloride IV on days 1 and 4, and vinorelbine ditartrate IV on day 1. Treatment repeats every 2-3 weeks for 2-3 courses in the absence of disease progression or unacceptable toxicity.
  * MOPP (mechlorethamine hydrochloride, vincristine, procarbazine hydrochloride, and prednisone): Patients receive MOPP combination chemotherapy comprising mechlorethamine hydrochloride IV on days 1 and 8, vincristine IV on days 1 and 8, oral procarbazine hydrochloride on days 1-14, and oral prednisone on days 1-14. Treatment repeats every 4 weeks for at least 2 courses in the absence of disease progression or unacceptable toxicity.

Patients with no progression of disease after salvage chemotherapy (at allograft work-up) proceed to allogeneic hematopoietic stem cell transplantation [AHSCT]* within 60 days after completion of salvage chemotherapy.

NOTE: *Patients with a nodal mass > 5 cm that has not ben previously irradiated and in the absence of extranodal disease may undergo involved-field radiotherapy twice daily for 2 weeks, prior to AHSCT.

* AHSCT with reduced-intensity or non-myeloablative conditioning: Patients achieving partial response or stable disease after salvage therapy receive fludarabine phosphate IV over 30 minutes on days -6 to -2; melphalan IV over 15 minutes on days -6 and -5; and undergo AHSCT on day 0 (reduced-intensity conditioning). Patients achieving complete response after salvage therapy receive fludarabine phosphate IV over 30 minutes on days -6 to -2; cyclophosphamide IV over 15 minutes on day -6; total-body irradiation over 20-30 minutes on day -1; and undergo AHSCT on day 0 (non-myeloablative conditioning).
* Graft-vs-host disease prophylaxis: Patients with related or unrelated donors receive cyclosporine IV over 2-4 hours or orally on days -3 to 100 followed by a taper, mycophenolate mofetil IV or orally on days -3 to 46 followed by a taper, and methotrexate IV on days 1, 3, 6, and 11.

Patients who received umbilical cord blood receive cyclosporine and mycophenolate mofetil as above (no methotrexate).

Follow-up period of 2 years post-transplant.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed classical Hodgkin lymphoma, including CD20+ disease

  * No lymphocyte predominant histology
* Primary refractory or relapsed disease with all 3 risk factors, failed platinum-based chemotherapy, or disease relapsed more than 100 days after autologous stem cell transplantation, proven by biopsy or fine-needle aspiration (cytology) of an involved site

  * Risk factors are defined as B-symptoms, extranodal sites of disease, and disease remission lasting < 1 year after first-line therapy
* Failed doxorubicin hydrochloride or mechlorethamine hydrochloride-containing front-line therapy
* Fludeoxyglucose F 18-PET scan demonstrating PET-avid disease
* No more than 2 prior salvage chemotherapy regimens (for patients proceed to allogeneic hematopoietic stem cell transplantation [AHSCT])
* Donor available meeting 1 of the following criteria (for patients proceed to AHSCT):

  * HLA-matched or one allele mismatched related donor

    * Genotypically or phenotypically matched at ≥ 9/10 of the A, B, C, DRB1, and DQB1 loci, as tested by high resolution
    * Peripheral blood stem cells (PBSC) collected
  * HLA-matched unrelated donor

    * Matched at ≥ 9/10 (allele mismatch only) of the A, B, C, DRB1, and DQB1 loci, as tested by high resolution
    * PBSC or bone marrow collected
  * Umbilical cord blood (2 units)

    * must be ≥ 4/6 HLA-A, B antigen, and DRB1 allele matched with recipient

PATIENT CHARACTERISTICS:

* Platelet count > 50,000/mm^3
* ANC > 1,000/mm^3
* Cardiac ejection fraction > 50% (for patients ≥ 18 years of age)
* Fractional shortening > 50% by echocardiogram* (for patients < 18 years of age)
* Adjusted diffusing capacity > 50% on pulmonary function testing*
* Serum creatinine < 1.5 mg/dL
* Creatinine clearance ≥ 50 mL/min
* Total bilirubin < 2.0 mg/dL in the absence of a history of Gilbert disease
* HIV I and II negative
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Karnofsky performance status (PS) ≥ 70% or Lansky PS ≥ 70% (for patients proceed to AHSCT)
* No active and uncontrolled infection at time of transplantation including active infection with Aspergillus or other mold (for patients proceed to AHSCT) NOTE: *measured since last chemotherapy

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior allogeneic transplantation
* No more than 1 prior autologous transplantation
* No inability to complete planned cytoreduction due to therapy complications

Ages: 13 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2007-11-13 (Actual); Primary Completion 2022-08-02 (Actual); Study Completion 2022-08-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Miguel-Angel Perales, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center; Juliet Barker, MBBS, Principal Investigator — Memorial Sloan Kettering Cancer Center; Tanya Trippett, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- High-Risk or Relapsed Hodgkin Lymphoma: This is a phase 2 intention-to-treat study of salvage chemotherapy followed by allogeneic HSC transplant for the treatment of primary refractory or relapsed HL. Patients who 1) do not progress on salvage chemotherapy, and 2) have both suitable HSC donors and 3) a satisfactory pre-allograft work-up will proceed to allograft. Patients who fail any of these 3 criteria will be off-study and considered treatment failures for the purposes of the intention-to-treat study.
  cyclophosphamide
  cyclosporine
  fludarabine phosphate
  gemcitabine hydrochloride
  ifosfamide
  mechlorethamine hydrochloride
  melphalan
  methotrexate
  mycophenolate mofetil
  prednisone
  procarbazine hydrochloride
  vincristine sulfate
  vinorelbine tartrate
  allogeneic bone marrow transplantation
  allogeneic hematopoietic stem cell transplantation
  nonmyeloablative allogeneic hematopoietic stem cell transplantation
  peripheral blood stem cell transplantation
  umbilical cord blood transplantation
  total-body irradiation
Period: Overall Study
Arm/Group | High-Risk or Relapsed Hodgkin Lymphoma
Started | 25
Completed | 24
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | High-Risk or Relapsed Hodgkin Lymphoma
Number analyzed (Participants) | 25
Age, Continuous [Median (Full Range); unit: years] | 35 [22 to 53]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 18
  Unknown or Not Reported | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 17
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival at 1 Year
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: 1 year
Measure: Number (95% Confidence Interval); unit: proportion of progression-free pts
Arm/Group | High-Risk or Relapsed Hodgkin Lymphoma
Number analyzed (Participants) | 24
proportion of progression-free pts | 33.3 [13 to 61.3]

2. Secondary Outcome: Overall Survival
Time Frame: up to 8 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | High-Risk or Relapsed Hodgkin Lymphoma
Number analyzed (Participants) | 24
months | 70.3 [51.5 to 96.1]

3. Secondary Outcome: Disease Relapse or Progression as Measured by CT Scan or PET
Time Frame: 3 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | High-Risk or Relapsed Hodgkin Lymphoma
Number analyzed (Participants) | 24
months | 34.3 [13.2 to 56.7]

ADVERSE EVENTS:
Time Frame: Up to 8 years
Arm/Group | High-Risk or Relapsed Hodgkin Lymphoma
All-Cause Mortality (participants affected / at risk) | 14/24
Serious Adverse Events (participants affected / at risk) | 6/24
Other Adverse Events (participants affected / at risk) | 2/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | High-Risk or Relapsed Hodgkin Lymphoma (N=24)
Death not assoc w CTCAE term - Death NOS (General disorders) | 2
Death not assoc w CTCAE term - Sudden Death (General disorders) | 1
Fatigue (General disorders) | 1
Fever (General disorders) | 1
Hematoma (Vascular disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | High-Risk or Relapsed Hodgkin Lymphoma (N=24)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-04): https://cdn.clinicaltrials.gov/large-docs/96/NCT00574496/Prot_SAP_000.pdf